CLINICAL TRIAL: NCT06020352
Title: Study on the Efficacy and Safety of KN046 Combined With Acitinib as a Neoadjuvant Therapy in Resectable Stage IB-IIIB Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: The Efficacy and Safety of KN046 Combined With Axitinib
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR003
Record Dates: First submitted 2023-08-23; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: NSCLC
Keywords: KN046; Axitinib; neoadjuvant
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): KN046 combined with axitinib as a neoadjuvant treatment regimen
  Interventions: Drug: KN046 plus Axitinib

INTERVENTIONS:
Drug: KN046 plus Axitinib — KN046 combined with axitinib as a neoadjuvant treatment regimen
  Other Names: surgical resection and selective adjuvant therapy with KN046

SUMMARY:
Evaluation of the efficacy of KN046 combined with acitinib as a neoadjuvant therapy for resectable NSCLC through primary pathological response rate and surgical resection rate

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the rate of major pathological remission (MPR) with preoperative use of KN046 versus axitinib, and thus to assess the efficacy of KN046 in combination with axitinib in patients with Stage IB-IIIB (Stage IIIB only T3N2M0) NSCLC (according to the 8th edition of the AJCC classification) who are scheduled to undergo surgery. Eligible subjects for this study were candidates for surgery for resectable stage IB-IIIB (stage IIIB only T3N2M0) NSCLC as judged by the investigator, with no evidence of distant metastases as assessed, and no evidence of unresectable local regional tumour extension.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years old and<75 years old on the day of signing the informed consent form, regardless of gender, and is willing to follow the research procedure;
2. Confirmed by histology or cytology as non-small cell lung cancer;
3. NSCLC patients evaluated by researchers as resectable in stage IB-IIIB (stage IIIB only limited to T3N2M0) (AJCC 8th edition);
4. Has not received any anti-tumor treatment in the past, including but not limited to systemic chemotherapy, immunotherapy, or radiotherapy;
5. No allergenic EGFR mutation or ALK change;
6. The ECOG score is 0-1 points.

Exclusion Criteria:

1. The lesion of squamous non-small cell lung cancer presents as a central type of lung cancer accompanied by cavity formation or invasion of blood vessels, with a high risk of hemoptysis;
2. Previously or currently suffering from interstitial pneumonia/lung disease that requires systemic hormone therapy;
3. Previous history of allogeneic bone marrow or organ transplantation;
4. Subjects who have undergone major surgical treatment (such as abdominal or thoracic surgery; excluding diagnostic puncture or peripheral vascular pathway replacement surgery) or have not recovered from surgical treatment within 28 days before the administration of this trial;
5. Prior to allocation, they have received systemic anti-cancer treatment, including research drugs targeting current malignant tumors;
6. Other known malignant tumors are progressing or require active treatment within the past 5 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (excluding bladder carcinoma in situ) who have received possible radical treatment are not excluded;
7. Pregnant and/or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
MPR | one month within postsurgery
  MPR is defined as the presence of ≤ 10% of active tumor cells in postoperative pathology (primary lesion).
Surgical resection rate | six weeks after last cycle of neoadjuvant therapy
  Surgical resection rate: refers to the proportion of subjects who completed the surgery according to the plan, defined as the distance from the last neoadjuvant treatment administration, and the surgical time ≤ 6 weeks.

SECONDARY OUTCOMES:
Complication rate | three months within postsurgery
  The incidence and severity of AE (classified according to CTCAE v5.0), severity, and their relationship with experimental treatment; Any abnormal results of laboratory tests, vital signs, and physical examinations;
pCR | one month within postsurgery
  PCR is defined as postoperative pathology (primary lesion) showing the absence of viable tumor cells
ORR | one month within postsurgery
  Defined as the proportion of subjects who achieved complete remission (CR) or partial remission (PR) according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: l: 2031222@tongji.edu.cn Chen, Dr, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No